CLINICAL TRIAL: NCT02534662
Title: A Prospective Study to Evaluate the Safety and Feasibility of an Endoluminal-suturing Device (Endomina TM) as an Aid for Endoscopic Gastric Reduction
Brief Title: Safety and Feasibility of an Endoluminal-suturing Device (Endomina TM) for Gastric Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mostafa Ibrahim, Gastroenterology and Hepatopancreatology Physician, Theodor Bilharz Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDOMINA
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Endomina will be introduced into the stomach over guide wires and then fixed to the endoscope. The procedure will include the placement of 4-6 transmural anterior-posterior sutures after argon plasma coagulation of the tissue opposition areas in order to ensure persistence of the pouch reduction. Patient will be kept overnight after the procedure.
  Interventions: Device: ENDOMINA

INTERVENTIONS:
Device: ENDOMINA — Endomina will be introduced into the stomach over guide wires and then fixed to the endoscope. The procedure will include the placement of 4-6 transmural anterior-posterior sutures after argon plasma coagulation of the tissue opposition areas in order to ensure persistence of the pouch reduction. Patient will be kept overnight after the procedure.

SUMMARY:
Objectives: Study to evaluate safety and feasibility of an endoluminal vertical gastroplasty (EVG) using an endoluminal-suturing device.

Briefly, Vertical gastric plication is a novel surgical approach for reducing the stomach capacity. Anterior surface plication and greater curvature plication are variations of vertical gastric plication that reduce the gastric capacity through infolding of the anterior surface or greater curvature of the stomach, respectively. These approaches have been tested, with positive results.

A transoral or endoluminal approach (ie, a procedure that requires no incision, because access is granted through the mouth) offers the potential for additional benefit to the patient, because the procedures continue to become more and more minimally invasive.

Advances in endoluminal devices are now allowing clinicians the ability to begin exploring bariatric procedures performed via flexible endoscopy. Although these procedures may not be as effective as their surgical counterparts, these less-invasive options may relieve patients of the significant risks associated with surgery.

Study duration and number of subjects A period of approximately 6 months is anticipated form the time the time the first patient is enrolled to the completion of the last patient.

The participants will be followed as follow:

Day (0): Procedure Day (+1): Clinical Follow up and discharge (i.e. if no adverse effects observed)

1 month: Follow up endoscopy, Clinical assessment 3 month: Follow up endoscopy, Clinical assessment 6 month: Final assessment (Endoscopically and Clinical) On Parallel a nutritional specialist will monitor the patient on quarterly basis (1,3,6,12).

Study procedures The intervention will be performed under general anesthesia with tracheal intubation. Endomina will be introduced into the stomach over guide wires and then fixed to the endoscope. The procedure will include the placement of 4-6 transmural anterior-posterior sutures after argon plasma coagulation of the tissue opposition areas in order to ensure persistence of the pouch reduction. Patient will be kept overnight after the procedure.

DETAILED DESCRIPTION:
Surgery is the only effective treatment for morbid obesity and can be divided into restrictive surgeries (Lap Band and Sleeve gastrectomy), malabsorptive surgeries (Biliary pancreatic deviation and duodenal switch) or a combination of both (RYGBP).

This later technique is the most common and most effective surgical procedure performed worldwide and has been processed to be an effective treatment of morbid obesity and its complications, achieving excess weight loss of 65 to 80 % ; 1-2 years after surgery.1 Vertical gastric plication is a novel surgical approach for reducing the stomach capacity. Anterior surface plication and greater curvature plication are variations of vertical gastric plication that reduce the gastric capacity through infolding of the anterior surface or greater curvature of the stomach, respectively. These approaches have been tested, with positive results. 3 A transoral or endoluminal approach (ie, a procedure that requires no incision, because access is granted through the mouth) offers the potential for additional benefit to the patient, because the procedures continue to become more and more minimally invasive.

Advances in endoluminal devices are now allowing clinicians the ability to begin exploring bariatric procedures performed via flexible endoscopy. Although these procedures may not be as effective as their surgical counterparts, these less-invasive options may relieve patients of the significant risks associated with surgery. 4

Endomina (Endo Tools Therapeutics, Nivelles, Belgium) is CE mark robot driven device that may be attached to an endoscope inside the body and allows remote manipulation of the arms of devices during a peroral intervention. It offers the possibilities of making transoral surgical full thickness sutures and may allow performing, via a transoral route.

Study design Prospective, non-randomized, open-label, single-center safety and feasibility study

Objectives:

Study to evaluate safety and feasibility of an endoluminal vertical gastroplasty (EVG) using an endoluminal-suturing device.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-64 years;
* BMI > 40 Kg/m2 or BMI >35 Kg/m2 with comorbidities
* Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: clinical assessment , endoscopy, radiography, as well as laboratory investigations.
* Must be able to understand and be willing to provide written informed consent.

Exclusion Criteria:

* Achalasia and any other esophageal motility disorders
* Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity.
* Hypertension: uncontrolled hypertension during last 3 month
* Severe renal, hepatic, pulmonary disease or cancer;
* GIT stenosis or obstruction
* Pregnancy or breastfeeding
* Impending gastric surgery 60 days post intervention;
* Currently participating in other study

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety characterized by the incidence of all Adverse Device Effects (ADEs), physical examination (vital signs), laboratory tests, and subsequent adverse events | 12 month
  Safety will be characterized by the incidence of all Adverse Device Effects (ADEs), non-serious and serious, possibly related to or related to the procedure and/or device that are experienced by study participants.
  In addition, safety assessments will be determined based on physical examination (vital signs) and laboratory tests during scheduled visits. Safety evaluations will also be performed to ensure no subsequent adverse events have occurred and to ensure any adverse events during the trial that are considered on-going are stable or have resolved. Safety will be assessed at 1 and 6 month following the intervention.

SECONDARY OUTCOMES:
Feasibility assessment obtained by measurements of total weight loss and excess weight loss | 12 month
  Information on efficacy will be obtained by measurements of total weight loss and excess weight loss during 6 month with an optional extension at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Deviere, PHD, Study Chair — Université Libre de Bruxelles
Locations (1):
- Erasme Hospital , ULB, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Huberty V, Ibrahim M, Hiernaux M, Chau A, Dugardeyn S, Deviere J. Safety and feasibility of an endoluminal-suturing device for endoscopic gastric reduction (with video). Gastrointest Endosc. 2017 Apr;85(4):833-837. doi: 10.1016/j.gie.2016.08.007. Epub 2016 Aug 22. PMID 27562938